CLINICAL TRIAL: NCT00282373
Title: Randomized Controlled Pilot Study: Induction of Mild Hypothermia in Resuscitated Cardiac Arrest Patients Using Traditional Surface Cooling Techniques vs. the Medivance® Arctic Sun® System
Brief Title: Induction of Mild Hypothermia in Resuscitated Cardiac Arrest Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medivance, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RESCUE
Record Dates: First submitted 2006-01-24; First posted 2006-01-26 (Estimated); Last update posted 2007-09-11 (Estimated); Status verified 2007-09

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest | interventions — Hypothermia, Induced

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: mild hypothermia

SUMMARY:
The primary objectives of this study are to determine the safety and feasibility of inducing mild hypothermia using a non-invasive thermoregulatory device, the Medivance Arctic Sun Temperature Management System, in patients resuscitated after cardiac arrest.

DETAILED DESCRIPTION:
Extensive research has been conducted in the use of mild hypothermia as a neuroprotectant in acute brain injury in animal models with studies having been initiated as far back as the 1950's. However, little work had been done in the area of therapeutic hypothermia and cardiac arrest.

In the early 80's, the Pittsburgh group resurrected the work with the induction of hypothermia in animals. The discovery of mild resuscitative hypothermia provided evidence that the main mechanism by which hypothermia can help resuscitate the brain after normothermic cardiac arrest is a synergistic effect of the suppression of deleterious chemical cascades, energy loss depolarization, calcium influx, excitotoxicity, free radical reactions, membrane failure, DNA fragmentation, and damage to the mitochondria).

Recently, the study "Mild hypothermia to improve the neurologic outcome after cardiac arrest" from the Hypothermia After Cardiac Arrest Study Group (New Engl J Med 2002;346:549-556) reported the results of a multicenter randomized controlled clinical trial that evaluated the effect of mild systemic hypothermia on mortality and functional outcome after resuscitation from out-of-hospital cardiac arrest due to ventricular fibrillation or tachycardia. Two hundred and seventy three patients were randomly assigned to standard normothermic or hypothermic management. Cooling to a target core body temperature of 32ºC to 34ºC was accomplished with the use of a specialized bed which delivers cold air over the entire body. Temperature was maintained in the target range for 24 hours after the start of cooling, followed by passive rewarming over 8 hours. Outcome was assessed at 6 months with a five point scale similar to the Glasgow Outcome Scale, dichotomized to classify independent patients with minimal or moderate disability to those who were dependent and severely disabled, vegetative, or dead. The results demonstrated a favorable neurological outcome in 55% of the 136 patients treated with hypothermia, compared to 39% of the 137 patients treated with normothermic management (risk ratio 1.40, 95% confidence interval 1.08 to 1.81, P=.009). . Mortality was also reduced with hypothermic management, from 41% in the hypothermia group to 55% in the normothermia group (risk ratio 0.74, 95% confidence interval 0.58 to 0.85, P=.02). In 19 patients (14%), the target temperature could not be reached. Complications did not differ significantly between the two groups, although there were trends toward increased rates of sepsis and bleeding with hypothermia.

Based upon the body of published evidence to date, the Advanced Life Support (ALS) Task Force of the International Liaison Committee on Resuscitation (ILCOR) made the following recommendations in October 2002 (Resuscitation 57 (2003) 231-235):

* Unconscious adult patients with spontaneous circulation after out-of-hospital cardiac arrest should be cooled to 32-34°C for 12 -24 hours when the initial rhythm is ventricular fibrillation (VF).
* Such cooling may also be beneficial for other rhythms or in-hospital cardiac arrest

The study is a prospective, randomized, multi-center, pilot study of the Arctic Sun System used as adjunctive therapy in patients resuscitated post cardiac arrest.

Patients who meet the inclusion criteria and for whom informed consent has been provided by an authorized representative/family member will be randomly assigned to either the control group (traditional cooling blankets and ice) or the experimental group (Arctic Sun Temperature Management System).

Patients will be cooled to a target range of 33.5°C to 33.9°C. The patient cooling will continue for 24 hours (from the initiation of cooling) and then gradually rewarmed to 36.0°C over approximately 6 to 12 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 18 years.
2. Witnessed out-of-hospital cardiac arrest of presumed cardiac origin in which the initial rhythm is ventricular fibrillation, ventricular tachycardia, pulseless electrical activity (PEA) or asystole.
3. First attempt at resuscitation (ACLS or CPR) by emergency medical personnel initiated within 15 minutes of collapse.
4. Restoration of spontaneous circulation (ROSC) within 60 minutes of collapse.
5. Time from restoration of spontaneous circulation to initiation of cooling is ≤ 6 hours.
6. Informed consent provided by authorized representative/family member.

Exclusion Criteria:

1. Temperature of less than 35C on admission.
2. Comatose or vegetative state prior to cardiac arrest.
3. Positive pregnancy test.
4. Purposeful response to verbal commands after ROSC and prior to initiation of hypothermia.
5. Evidence of hypotension (MAP<60) for more than 30 minutes after ROSC and prior to initiation of hypothermia.
6. Evidence of hypoxia (oxygen saturation<85% despite supplemental oxygen) for more than 15 minutes after ROSC and prior to initiation of hypothermia.
7. Terminal illness that preceded the arrest (life expenctancy < 1 year).
8. Patients experiencing cardiogenic shock.
9. Patients continuing to experience refractory ventricular arrhythmias at the time of enrollment.
10. Patients receiving 2 or more high dose vasopressors.
11. Active bleeding or known preexisting coagulapathy.
12. Patient history of cold agglutinin disease.
13. Patient history of Raynaud's Disease.
14. Patient history of Sickle Cell disease.
15. Evidence of compromised skin integrity or irregularities (such as urticaria, rash, lacerations, burns, abrasions.
16. Patient weight > 114 kg (250 lbs) or < 50 kg (110 lbs)
17. Enrollment in another therapeutic study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2004-11; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Feasibility -patient temperature below 34C within 4 hours
Feasibility -maintain patient target temperature for 24 hrs
Safety - serious adverse events, mortality

SECONDARY OUTCOMES:
Effectiveness - neurological outcome measured by OPC/CPC

CONTACTS AND LOCATIONS:
Overall Officials: Kennon Heard, M.D., Principal Investigator — University of Colorado, Denver
Locations (6):
- United States (6):
  - University of Arizona Medical Center, Tucson, Arizona
  - University of Colorado Health Science Center, Denver, Colorado
  - Johns Hopkins - Bayview Medical Center, Baltimore, Maryland
  - William Beaumont Hospital, Royal Oak, Michigan
  - Ohio State University Medical Center, Columbus, Ohio
  - Virginia Commonwealth University Medical Center, Richmond, Virginia

REFERENCES:
- [Derived] Heard KJ, Peberdy MA, Sayre MR, Sanders A, Geocadin RG, Dixon SR, Larabee TM, Hiller K, Fiorello A, Paradis NA, O'Neil BJ. A randomized controlled trial comparing the Arctic Sun to standard cooling for induction of hypothermia after cardiac arrest. Resuscitation. 2010 Jan;81(1):9-14. doi: 10.1016/j.resuscitation.2009.09.015. Epub 2009 Oct 24. PMID 19854555